CLINICAL TRIAL: NCT02302508
Title: PANDDA Study: Pharmacokinetics of Antiplatelet Drugs in Diabetic pAtients
Brief Title: Pharmacokinetics of Antiplatelet Drugs in Diabetic pAtients
Acronym: PANDDA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14.143
Record Dates: First submitted 2014-11-11; First posted 2014-11-27 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2017-08

CONDITIONS: Diabetes
Keywords: pharmacokinetics; drug metabolism; platelet reactivity; carboxylesterase; cytochromes p450; type 2 diabetes; active metabolite
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T2D patients with A1C ≤7.0 (Experimental): Clopidogrel, Prasugrel, Ticagrelor A single oral dose of clopidogrel 300 mg or prasugrel 60 mg or ticagrelor 180 mg in a randomized fashion on 3 different occasions (washout period of 12 days or more)
  Interventions: Drug: Clopidogrel, Prasugrel, Ticagrelor
- T2D patients with A1C>7.5 (Experimental): Clopidogrel, Prasugrel, Ticagrelor A single oral dose of clopidogrel 300 mg or prasugrel 60 mg or ticagrelor 180 mg in a randomized fashion on 3 different occasions (washout period of 12 days or more)
  Interventions: Drug: Clopidogrel, Prasugrel, Ticagrelor
- Insulino-treated (Experimental): Clopidogrel, Prasugrel, Ticagrelor A single oral dose of clopidogrel 300 mg or prasugrel 60 mg or ticagrelor 180 mg in a randomized fashion on 3 different occasions (washout period of 12 days or more)
  Interventions: Drug: Clopidogrel, Prasugrel, Ticagrelor
- Non-diabetic healthy subjects (Active Comparator): Clopidogrel, Prasugrel, Ticagrelor A single oral dose of clopidogrel 300 mg or prasugrel 60 mg or ticagrelor 180 mg in a randomized fashion on 3 different occasions (washout period of 12 days or more)
  Interventions: Drug: Clopidogrel, Prasugrel, Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel, Prasugrel, Ticagrelor — PK and PD parameters will be compared between groups and comparison will be performed between antiplatelet agents
  Other Names: Plavix; Brilinta; Effient

SUMMARY:
Clopidogrel efficacy appears diminished in patients with type 2 diabetes (T2D) who continue to show an increased risk of adverse cardiovascular events and mortality compared to those without T2D.The aim of the first project is to describe the pharmacokinetic (PK) profile of three antiplatelet drugs in 4 groups of patients according to their diabetic or non-diabetic status. To this end, PK profiles will be determined after a single oral dose of 300 mg clopidogrel, 60 mg prasugrel and 180 mg ticagrelor in patients (n=108); 1) with T2D and good glycemic control; 2) with T2D and poor glycemic control; 3) with insulin-treated diabetes; and 4) non-diabetic subjects.

DETAILED DESCRIPTION:
Clopidogrel efficacy appears diminished in patients with T2D who continue to show an increased risk of adverse cardiovascular events and mortality compared to those without T2D. To the contrary, response to prasugrel and ticagrelor appears conserved in ACS patients with diabetes. There are several mechanisms that may be contributing to the blunted response to clopidogrel but a postulated decreased concentration of clopidogrel active metabolite is worth pursuing further.

The overall objective of this proposal is to describe the pharmacokinetic profiles of three antiplatelet drugs namely, clopidogrel, prasugrel and ticagrelor in four groups of patients according to their diabetic or non-diabetic status.

Patients (n=108) will be recruited to constitute 4 groups: Group I, 27 confirmed T2D with A1C ≤7; Group II, 27 patients with poor glycemic control A1C Patients (n=108) will be recruited to constitute 4 groups: Group I, 27 confirmed T2D with A1C <7.0; Group II, 27 patients with poor glycemic control A1C >7.5; Group III, 27 patients with insulin-treated T2D; and Group IV, 27 sex-matched non-diabetic healthy subjects. Subjects with type 2 diabetes according to the Canadian Clinical Guidelines will be recruited at the CHUM outpatient clinic. After an overnight fast, participants will be admitted to the CRCHUM's Clinical Research Unit (they will not be hospitalized). A crossover randomized study design with 3 phases (washout period of 12 days between phases) will be conducted. Subjects will receive a single oral dose of clopidogrel 300 mg or prasugrel 60 mg or ticagrelor 180 mg in a randomized fashion on 3 different occasions. Serial blood samples will be drawn and urine collected over 10 hours (PK and PD analysis).

A blood sample will be taken for pharmacogenetic analyses. Additional blood samples will be collected just before the administration of antiplatelet drugs to measure fasting insulin, glycaemia levels to determine the HOMA-IR. In addition, the following covariates namely, gender, age, weight, duration of diabetes and drug profile will be also recorded.

Their regular medication will be administered 4 hours after the administration of the antiplatelet drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥18 years old
* Non-smokers (>3 months)
* T2D with good glycemic control A1C<7.0
* T2D with poor glycemic control A1C >7.5
* Insulin-treated T2D
* Non-diabetic healthy subjects

Exclusion Criteria:

* Subjects with estimated glomerular filtration (MDRD) <50 mL/min/1.73m2
* ALT and AST 3 times above the upper limit of normal
* Organ transplant recipients
* Inflammatory illnesses (i.e., polyarthritis, hepatitis, cirrhosis, active infectious diseases)
* Active cancer (except non-melanoma skin cancer)
* Uncontrolled thyroid functions
* Inflammatory bowel diseases (ulcerous colitis and Crohn's disease), bariatric surgery
* Pregnancy
* History of drug or alcohol abuse
* Platelet function disorder,
* One of the following therapies : P2Y12 inhibitors, antithrombotics, antibiotics, anticoagulant, antivirals, CYP450 inducers (carbamazepine, phenobarbital, phenytoin, rifampin, St-John's worth), CYP450 inhibitors (amiodarone, fluoxetine, verapamil), immunosuppressors, INFs, or grapefruit juice (<4 weeks) or an investigational drug
* Intolerance or hypersensitivity to antiplatelet drugs or their excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC0-t metabolites and parent drug) of clopidogrel, prasugrel and ticagrelor. | 30 days
  The association between the T2D effects on antiplatelet drug's PK (AUC0-t metabolites, AUC0-t of parent drug) will be assessed after a single oral loading dose in patients with different diabetic status.

SECONDARY OUTCOMES:
Platelet function activities | 30 days
  Platelet function reactivity (pharmacodynamic) will be compared between antiplatelet agents and groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, BPharm. PhD, Principal Investigator — Centre de recherche du Centre Hospitalier de l'université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada